CLINICAL TRIAL: NCT00943137
Title: The Optimisation of 5-Fluorouracil Dose by Pharmacokinetic Monitoring in Asian Patients With Advanced Stage Cancer
Brief Title: The Optimization of 5-Fluorouracil Dose by Pharmacokinetic Monitoring in Asian Patients With Advanced Stage Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK01/06/09
Record Dates: First submitted 2009-07-16; First posted 2009-07-22 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Cancer (Advanced Stage)
MeSH Terms: conditions — Neoplasms | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-FU dosage adjustments (Experimental): The dose of continuous infusion 5-FU will be adjusted every cycle until patients reached the therapeutic plasma range (450 to 550 microgram/L).
  Interventions: Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: 5-Fluorouracil — Chemotherapy will be one of the following:
  1. de Gramont: folinic acid 400mg/m2 day 1, 5-FU 400 mg/m2 bolus on day 1 followed by 46 hour continuous infusion of 5-FU 2400mg/m2.
  2. FOLFIRI: Irinotecan 180mg/m2 on day 1, folinic acid 400mg/m2 day 1, 5-FU 400 mg/m2 bolus on day 1 followed by 46 hour continuous infusion of 5-FU 2400mg/m2.
  3. Modified FOLFOX-6: Oxaliplatin 85mg/m2 on day 1, folinic acid 400mg/m2 day 1, 5-FU 400 mg/m2 bolus on day 1 followed by 46 hour continuous infusion of 5-FU 2400mg/m2.

SUMMARY:
The purpose of this study is:

1. To determine the proportion of Asian patients achieving a target area under the curve (AUC) of 20-24 mg.h/L using a pharmacokinetically guided 5-fluorouracil (5-FU) dose
2. To determine the safety and tolerability of dose adjusted 5-FU
3. To correlate 5-FU pharmacokinetics with gene variants associated with the 5-FU pathway and with clinical outcomes

Based on Western data, levels of 5-FU are highly variable when doses are based on BSA. A relationship between systemic plasma levels of 5-FU and treatment toxicity and efficacy exists. Whilst pharmacokinetically-guided dose management has been shown to improve 5-FU efficacy and tolerance, there is currently no data in Asian patients using this approach. Using pharmacokinetically guided 5-FU-dose adjustment, the investigators hypothesize the proportion of Asian patients achieving a target AUC of 20-24 mg.h/L is similar to that of Caucasians.

METHODS:

This is an open, non-randomised single center Phase II study evaluating dose adjusted 5-FU in patients receiving de Gramont, FOLFIRI or mFOLFOX-6 schedules.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged = 21 years to 80 years
* Histologically proven advanced stage carcinoma where De Gramont, FOLFIRI or mFOLFOX-6 regimen is indicated.
* No more than one line of prior chemotherapy for advanced stage disease
* Measurable disease according to RECIST criteria or evaluable disease
* Karnofsky performance status of at least 70% or electrocorticogram performance status ? 2
* A life expectancy of at least 3 months
* absolute neutrophil count > 1.5 x 10^9/L
* Platelet count > 100 x 10^9/L.
* Total bilirubin > 1.5x upper limits of normal reference range (ULN)
* AST/ALT levels > 2.5x upper limit of normal. If hepatic metastases are present, these parameters could be ? 5x the ULN.
* Women of reproductive age and men must agree to practice effective contraception during the entire study period. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-child-bearing potential. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Signed informed consent

Exclusion Criteria:

* Received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, biologic or any investigational therapy within 21 days prior to study drug administration (6 weeks for mitomycin or nitroureas) and have not recovered from therapy.
* Patients who have not recovered from major surgery
* Subjects with treated brain metastases are eligible provided they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to study drug administration).
* Clinically significant cardiac disease, e.g. myocardial infarction within the last 12 months.
* Known HIV infection
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, other serious uncontrolled concomitant disease, psychiatric illness/ social situation that would limit study compliance.
* Known allergies to any component of the drug regime
* Organ allografts
* Known dihydropyrimidine dehydrogenase deficiency

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2009-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
AUC of 20-24 mg.h/L | 28 days - 2 cycles
  If patient achieved target AUC for two consecutive cycles, therapeutic dose monitoring will performed every alternate cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Soh, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Meta-analysis Group In Cancer; Piedbois P, Rougier P, Buyse M, Pignon J, Ryan L, Hansen R, Zee B, Weinerman B, Pater J, Leichman C, Macdonald J, Benedetti J, Lokich J, Fryer J, Brufman G, Isacson R, Laplanche A, Levy E. Efficacy of intravenous continuous infusion of fluorouracil compared with bolus administration in advanced colorectal cancer. J Clin Oncol. 1998 Jan;16(1):301-8. doi: 10.1200/JCO.1998.16.1.301. PMID 9440757
- [Background] Meta-Analysis Group In Cancer; Levy E, Piedbois P, Buyse M, Pignon JP, Rougier P, Ryan L, Hansen R, Zee B, Weinerman B, Pater J, Leichman C, Macdonald J, Benedetti J, Lokich J, Fryer J, Brufman G, Isacson R, Laplanche A, Quinaux E, Thirion P. Toxicity of fluorouracil in patients with advanced colorectal cancer: effect of administration schedule and prognostic factors. J Clin Oncol. 1998 Nov;16(11):3537-41. doi: 10.1200/JCO.1998.16.11.3537. PMID 9817272